CLINICAL TRIAL: NCT01552187
Title: COlchicine for Prevention of the Post-pericardiotomy Syndrome and Post-operative Atrial Fibrillation (COPPS-2 Trial).
Acronym: COPPS-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maria Vittoria Hospital (Other)
Responsible Party: Principal Investigator, Massimo Imazio, Principal Investigator, Maria Vittoria Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 86/19/11; 2011-005835-21 (EudraCT Number)
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Cardiac Surgery; Post-pericardiotomy Syndrome; Atrial Fibrillation; Pericardial Effusion; Pleural Effusion
Keywords: cardiac surgery; post-pericardiotomy syndrome; atrial fibrillation; pericardial effusion; pleural effusion; prevention; colchicine
MeSH Terms: conditions — Postpericardiotomy Syndrome; Atrial Fibrillation; Pericardial Effusion; Pleural Effusion | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Colchicine (Active Comparator): Colchicine
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5 mg BID or colchicine 0.5mg (<70kg) 48 to 72 hours before surgery till 1 months after surgery
  Arms: Colchicine
Drug: Placebo — Placebo 48 to 72 hours before surgery till 1 months after surgery
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized trial to assess the efficacy and safety of colchicine for post-pericardiotomy syndrome prevention, post-operative effusions prevention, and post-operative atrial fibrillation prevention.

DETAILED DESCRIPTION:
This is a multi center, double-blind, randomized trial to test the efficacy and safety of colchicine for prevention of post-pericardiotomy syndrome, post-operative effusions, and post-operative atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18years
* Candidate to cardiac surgery but cardiac transplantation
* Informed consent

Exclusion Criteria:

* Atrial fibrillation
* Candidate to cardiac transplantation
* Severe liver disease or elevation of serum transaminases (> 1.5 times the upper reference limit)
* Serum creatinine > 2.5 mg/dL
* Preoperative elevation of CK or known myopathy
* Known chronic intestinal diseases or blood dyscrasias
* Pregnancy, Lactation or Women of childbearing potential not protected by a contraception method
* Hypersensitivity to colchicine
* Treatment with colchicine for any cause

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Post-pericardiotomy syndrome, post-operative effusions, post-operative atrial fibrillation incidence | 3 months
  Incidence of the outcomes at 3 months from cardiac surgery

SECONDARY OUTCOMES:
Cardiac Tamponade or Need for Pericardiocentesis | 3 months
Need for thoracentesis | 3 months
Recurrence of the post-pericardiotomy syndrome | 3 months
Re-admission | 3 months
Overall mortality | 3 months
Stroke incidence | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Dpt. Maria Vittoria Hospital, Torino, Torino, Italy

REFERENCES:
- [Derived] Imazio M, Brucato A, Ferrazzi P, Pullara A, Adler Y, Barosi A, Caforio AL, Cemin R, Chirillo F, Comoglio C, Cugola D, Cumetti D, Dyrda O, Ferrua S, Finkelstein Y, Flocco R, Gandino A, Hoit B, Innocente F, Maestroni S, Musumeci F, Oh J, Pergolini A, Polizzi V, Ristic A, Simon C, Spodick DH, Tarzia V, Trimboli S, Valenti A, Belli R, Gaita F; COPPS-2 Investigators. Colchicine for prevention of postpericardiotomy syndrome and postoperative atrial fibrillation: the COPPS-2 randomized clinical trial. JAMA. 2014 Sep 10;312(10):1016-23. doi: 10.1001/jama.2014.11026. PMID 25172965
- [Derived] Imazio M, Belli R, Brucato A, Ferrazzi P, Patrini D, Martinelli L, Polizzi V, Cemin R, Leggieri A, Caforio AL, Finkelstein Y, Hoit B, Maisch B, Mayosi BM, Oh JK, Ristic AD, Seferovic P, Spodick DH, Adler Y. Rationale and design of the COlchicine for Prevention of the Post-pericardiotomy Syndrome and Post-operative Atrial Fibrillation (COPPS-2 trial): a randomized, placebo-controlled, multicenter study on the use of colchicine for the primary prevention of the postpericardiotomy syndrome, postoperative effusions, and postoperative atrial fibrillation. Am Heart J. 2013 Jul;166(1):13-9. doi: 10.1016/j.ahj.2013.03.025. Epub 2013 May 6. PMID 23816016